CLINICAL TRIAL: NCT05571826
Title: Effectiveness of Telerehabilitation Interventions in Persons With Multiple Sclerosis: Patient Perspective
Brief Title: Effectiveness of Telerehabilitation Interventions in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Serkan Ozakbas, MD, Dokuz Eylul University
Other Study IDs: 7409-GOA
Record Dates: First submitted 2022-10-06; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; upper extremity; telerehabilitation; patient perspective
MeSH Terms: conditions — Multiple Sclerosis | interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- telerehabilitation: Assessments, no specific intervention
  Interventions: Behavioral: telerehabilitation

INTERVENTIONS:
Behavioral: telerehabilitation — No specific treatments will be applied. The persons who experienced telerehabilitation interventions will be included.

SUMMARY:
Multiple sclerosis (MS) is an inflammatory, demyelinating, neurodegenerative disease of the central nervous system of unknown etiology. The most common clinical signs and symptoms are motor dysfunction, fatigue, spasticity, impaired mobility, cognitive impairment, chronic pain, depression, decreased quality of life, and bladder and bowel dysfunction. 66% of people with MS have impaired upper extremity function. As a result of the deterioration in upper extremity function, the performance of many daily living activities affects performance. As a result of this influence, there is a decrease in the functional independence of people, quality of life, and participation in activities in the community. Exercise training represents an existing behavioral treatment approach to safely manage many functional, symptomatic, and quality-of-life outcomes in MS. Telerehabilitation has been defined as "the delivery of rehabilitation services through information and communication technologies." Telerehabilitation has proven to be useful for people with MS by increasing physical activity and reducing fatigue. In the studies, telerehabilitation and face-to-face rehabilitation services were compared, and stated that they had similar results. At the same time, it was stated that telerehabilitation provides people with gains in terms of time and cost. In addition to all these, the researchers emphasized the benefits they received from telerehabilitation from the people's statements. Therefore, the results of this study, which will be performed on MS patients, will enable the evaluation of telerehabilitation strategies from the patient's point of view.

The participants was included in the study titled 'Investigation of the Effects of the Synchronized Telerehabilitation-based Upper Extremity Training Program on Hand-arm Function, Pain, Fatigue, Quality of Life, and Participation in People With Multiple Sclerosis (ClinicalTrials.gov Identifier: NCT05073731)' will be included in this study. Questionnaires that will enable individuals to evaluate their telerehabilitation service will be administered once. Physicians and physiotherapists will make evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Having a definitive diagnosis of MS according to the 2017 McDonald criteria
* Being over 18 years old
* Volunteering to participate in the study
* To have received exercise training based on synchronous or asynchronous telerehabilitation

Exclusion Criteria:

* Having a neurological disease other than MS
* Having an MS attack 30 days before or during the study
* Cognitive disability at a level that hinders assessment and treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The people with multiple sclerosis who have received exercise training based on synchronous or asynchronous telerehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Telehealth Usability Questionnaire | Baseline
  Telehealth Usability Questionnaire was developed by Bakken et al. in 2006. The 21-item questionnaire evaluated the satisfaction and usability of people receiving telemedicine services. A 5-item Likert scale is used in the evaluation. The total score ranges from 21 to 105. Turkish validity and reliability were established.
Telemedicine Satisfaction Questionnaire | Baseline
  Demiris et al. Developed by It consist of 17 items in total. A 5-item Likert-type scale is used to evaluate telemedicine service, expectation, satisfaction, and usability of people. The total score is scored between 17 and 85. Turkish validity and reliability were established.

SECONDARY OUTCOMES:
Expanded Disability Status Scale | Baseline
  Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The Expanded Disability Status Scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Ozakbas, MD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided